CLINICAL TRIAL: NCT00416494
Title: Phase II Study of Oxaliplatin, Capecitabine and Bevacizumab in the Treatment of Metastatic Colorectal Cancer
Brief Title: Capecitabine, Oxaliplatin, and Bevacizumab in Treating Patients With Metastatic or Recurrent Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Hurwitz, MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008646; DUMC-4951-05-7R2; GENENTECH-DUMC-4951-05-7R2; SANOFI-DUMC-4951-05-7R2; ROCHE-DUMC-4951-05-7R2; CDR0000449971 (Other: NCI)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

ARMS (2):
- Initial Cohort (Experimental)
  Interventions: Biological: bevacizumab; Drug: oxaliplatin; Drug: Capecitabine
- Second cohort (Experimental)
  Interventions: Biological: bevacizumab; Drug: oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Biological: bevacizumab — 10 mg/kg intravenously over 30-90 minutes on day 1
Drug: oxaliplatin — 85 mg/m2 intravenously over 2 hours on day 1.
Drug: Capecitabine — Oral administration every 12 hours on days 1-5 and 8-12 1000 mg/m2 in initial cohort
  Arms: Initial Cohort
Drug: Capecitabine — Oral administration every 12 hours on days 1-5 and 8-12 850 mg/m2 in second cohort
  Arms: Second cohort

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving capecitabine and oxaliplatin together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving oxaliplatin and capecitabine together with bevacizumab works in treating patients with metastatic or recurrent colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the response rate in patients with previously untreated metastatic colorectal cancer treated with capecitabine, oxaliplatin, and bevacizumab.

Secondary

* Assess time to progression (TTP), disease-free survival (DFS), and overall survival (OS) in patients treated with this regimen.
* Assess the safety and tolerability of bevacizumab, oxaliplatin, and capecitabine in patients with previously untreated metastatic colorectal cancer.

Exploratory

* Evaluate the effect of this regimen on the biomarkers of angiogenesis.
* Assess the effect of this regimen on wound angiogenesis.

OUTLINE: Patients receive oral capecitabine twice daily on days 1-5 and 8-12, oxaliplatin IV over 2 hours on day 1, and bevacizumab IV over 1-1½ hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically documented adenocarcinoma of the colon or rectum

  * Metastatic or recurrent disease not amenable to potentially curative treatment (e.g., inoperable metastatic disease)
* No leptomeningeal or brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* AST/ALT < 2.5 times upper limit of normal (ULN) (5 times ULN if known liver metastases)
* Bilirubin < 1.5 times ULN
* Creatinine clearance > 50 mL/min
* No unstable or poorly controlled hypertension (> 150/100 mm Hg)

  * Patients who have recently started or adjusted antihypertensive medications are eligible provided blood pressure is < 140/90 mm Hg on any new regimen for at least 3 different observations over 14 days
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study and for at least 3-4 months after study completion
* No arterial or venous thrombosis (including cerebrovascular accident) within the last 3 months
* No known, existing, uncontrolled coagulopathy
* No clinically significant cardiac disease
* No congestive heart failure
* No symptomatic coronary artery disease
* No cardiac arrhythmias not well controlled with medication
* No myocardial infarction within the last 12 months
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to oxaliplatin, capecitabine, or bevacizumab
* No history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk from treatment complications

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior sorivudine or brivudine
* At least 6 months since prior adjuvant treatment with fluorouracil and leucovorin calcium or a fluorouracil and leucovorin calcium-based regimen
* No major surgery within 4 weeks without complete recovery
* No prior chemotherapy for metastatic/recurrent disease
* No cancer immunotherapy or other biologic therapy while on therapy
* No radiotherapy while on study
* No hormonal therapy for cancer while on study
* No full-dose warfarin (INR of > 1.5), heparin (> 10,000 units/day), or thrombolytic agents
* Allopurinol and cimetidine should be discontinued prior to starting on this regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-09; Primary Completion 2008-01 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I. Hurwitz, MD, Principal Investigator — Duke Cancer Institute

REFERENCES:
- [Result] Hurwitz H, Fernando N, Yu D, et al.: A phase II study of oxaliplatin, capecitabine and bevacizumab in the treatment of metastatic colorectal cancer. [Abstract] Ann Oncol 16 (Suppl 2): A-55P, ii285, 2005.
- [Derived] Liu Y, Starr MD, Bulusu A, Pang H, Wong NS, Honeycutt W, Amara A, Hurwitz HI, Nixon AB. Correlation of angiogenic biomarker signatures with clinical outcomes in metastatic colorectal cancer patients receiving capecitabine, oxaliplatin, and bevacizumab. Cancer Med. 2013 Apr;2(2):234-42. doi: 10.1002/cam4.71. Epub 2013 Mar 6. PMID 23634291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited between September 2003 and July 2005 in the Duke Cancer Center and Duke Oncology Network sites.
Groups:
- Initial Cohort: oxaliplatin : 85 mg/m2 intravenously over 2 hours on day 1.
  Capecitabine : Oral administration every 12 hours on days 1-5 and 8-12 1000 mg/m2 in initial cohort
  bevacizumab : 10 mg/kg intravenously over 30-90 minutes on day 1
- Second Cohort: oxaliplatin : 85 mg/m2 intravenously over 2 hours on day 1.
  bevacizumab : 10 mg/kg intravenously over 30-90 minutes on day 1
  Capecitabine : Oral administration every 12 hours on days 1-5 and 8-12 850 mg/m2 in second cohort
Period: Overall Study
Arm/Group | Initial Cohort | Second Cohort
Started | 19 | 31
Completed | 19 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Cohort | Second Cohort | Total
Number analyzed (Participants) | 19 | 31 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 26 | 40
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (13.3) | 55.3 (12.6) | 55 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 18 | 23
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 19 | 31 | 50

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Percentage of Participants With Partial or Complete Response)
Description: Restaging scans occurred every 9 weeks from time of study drug initiation until disease progression.
  Disease assessment was performed and recorded according to the Response Evaluation Criteria in Solid Tumors (RECIST v.1.0) Guidelines.
  The definitions were:
  Complete response (CR)- Disappearance of all target lesions Partial response (PD)- At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Stable disease (SD)- Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Progressive disease (PD) - At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: After all subjects were evaluated for restaging which occured every 9 weeks from drug initiation until disease progression, assesed up to 24 months.
Population: All subjects who had restaging scans were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants with response
Arm/Group | Initial Cohort | Second Cohort
Number analyzed (Participants) | 19 | 31
percentage of participants with response | 63 [38 to 84] | 42 [25 to 61]

2. Secondary Outcome: Time to Progression
Description: Disease assessment was performed and recorded according to the Response Evaluation Criteria in Solid Tumors (RECIST v.1.0) Guidelines.
  Progressive disease is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: From time of treatment until documented progression, assesed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Cohort | Second Cohort
Number analyzed (Participants) | 19 | 31
months | 10.1 (5.7) [5.7 to 19.5] | 10.4 [6.9 to 15.4]

3. Secondary Outcome: Disease Free Survival
Description: as for outcome 2
Time Frame: From time of treatment until documented progression or death from any cause, whichever came first, assesed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Cohort | Second Cohort
Number analyzed (Participants) | 19 | 31
months | 10.1 [5.7 to 19.5] | 10.4 [6.9 to 15.4]

4. Secondary Outcome: Overall Survival
Description: Average months of survival of participants after receiving study drug.
Time Frame: From time of treatment until death from any cause, assesed up to 60 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Cohort | Second Cohort
Number analyzed (Participants) | 19 | 31
months | 19.6 [13.3 to 30.2] | 24.8 [12.9 to 39.7]

5. Secondary Outcome: Safety and Tolerability
Description: Number of participants with adverse events
Time Frame: After all participants went off study drug regimine.
Measure: Number; unit: participants with adverse event
Arm/Group | Initial Cohort | Second Cohort
Number analyzed (Participants) | 19 | 31
participants with adverse event | 19 | 29

6. Other Pre Specified Outcome: Effect on Angiogenesis Biomarkers
Time Frame: After study completion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Effect on Wound Angiogenesis
Time Frame: After study completion
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Initial Cohort | Second Cohort
Serious Adverse Events (participants affected / at risk) | 6/19 | 9/31
Other Adverse Events (participants affected / at risk) | 19/19 | 29/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Cohort (N=19) | Second Cohort (N=31)
Bowel Perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute Calculus Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Wound Dehisence (General disorders) | 1 (1) | 0 (0)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 0 (0) | 1 (1)
Altered mental status (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Angina (Cardiac disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Cohort (N=19) | Second Cohort (N=31)
Anorexia (Gastrointestinal disorders) | 15 (15) | 17 (17)
Abdominal Cramping (Gastrointestinal disorders) | 8 (8) | 12 (12)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 4 (4)
Neutropenia (Investigations) | 4 (4) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (11) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 10 (10)
Dehydration (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 16 (16) | 20 (20)
Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 16 (16) | 23 (23)
Fever (General disorders) | 4 (4) | 3 (3)
Flatuance (Gastrointestinal disorders) | 0 (0) | 3 (3)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 15 (15) | 11 (11)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Infection (Infections and infestations) | 4 (4) | 2 (2)
Insomnia (General disorders) | 12 (12) | 12 (12)
Nausea (Gastrointestinal disorders) | 14 (14) | 16 (16)
Pain (General disorders) | 13 (13) | 20 (20)
Skin rash (Skin and subcutaneous tissue disorders) | 14 (14) | 16 (16)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Vomiting (Gastrointestinal disorders) | 8 (8) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No